CLINICAL TRIAL: NCT04720456
Title: Noninvasive Subharmonic Aided Pressure Estimation of Portal Hypertension in Children
Brief Title: SHAPE of Portal Hypertension in Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Children's Hospital of Philadelphia (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20F.728; R01DK118964 (NIH)
Record Dates: First submitted 2021-01-04; First posted 2021-01-22 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Hypertension, Portal
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Intervention Model Description: A prospective randomized cohort study with a longitudinal arm. There will be 2 cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- SHAPE with Sonazoid (Experimental): Up to 60 children (6-21 years of age) with a diagnosis of chronic liver disease, including some who will have portal hypertension who are followed at The Children's Hospital of Philadelphia (CHOP) will be enrolled in this arm. A SHAPE measurement using the ultrasound contrast agent Sonazoid® (perfluorobutane microbubbles) will be performed during a single visit. A dose of three vials with 16 μL each of microbubbles will be prepared. An infusion of the ultrasound contrast agent at the rate of 0.18 mL/kg/hour will be co-infused with an infusion of saline at the rate of 120 mL/hour resulting in an effective dosage of 1.44 μL microbubbles/kg/hour as per the FDA approved IND through an IV line in a peripheral vein. The total duration of contrast agent infusion is expected to range from 4 to 8 minutes, which includes a 2 min calibration period followed by 2-6 minutes of SHAPE acquisition (i.e., ultrasound imaging).
  Interventions: Drug: SHAPE measurement using the ultrasound contrast agent Sonazoid (perfluorobutane microbubbles)
- SHAPE with Lumason (Active Comparator): Up to 60 children (6-21 years of age) with a diagnosis of chronic liver disease, including some who will have portal hypertension who are followed at CHOP will be enrolled in this arm. A SHAPE measurement using the ultrasound contrast agent LUMASON® (sulfur hexafluoride lipid-type A microspheres) will be performed during a single visit. Two doses of 0.03 mL/kg (or 2.4 mL maximum) as per package labeling will be prepared and mixed with saline at a 1:10 dilution in a 50 ml bag of saline. The diluted preparation of Lumason will be through an IV line in a peripheral vein up to 4 mL/min using an infusion setup. The total duration of contrast agent infusion is expected to range from 4 to 8 minutes, which includes a 2 min calibration period followed by 2-6 minutes of SHAPE acquisition (i.e., ultrasound imaging).
  Interventions: Drug: SHAPE measurement using the ultrasound contrast agent Lumason (sulfur hexafluoride lipid-type A microspheres)
- Longitudinal SHAPE (Experimental): SHAPE will be used to monitor subjects identified in the initial examination as having portal hypertension for up to 18 months. These subjects will undergo laboratory testing every 6 months as a part of their clinical standard of care. During these times the SHAPE examination will also be repeated using the same ultrasound contrast agent and infusion methodologies (including dosages) as during the initial study.
  Interventions: Drug: SHAPE measurement using the ultrasound contrast agent Sonazoid (perfluorobutane microbubbles); Drug: SHAPE measurement using the ultrasound contrast agent Lumason (sulfur hexafluoride lipid-type A microspheres)

INTERVENTIONS:
Drug: SHAPE measurement using the ultrasound contrast agent Sonazoid (perfluorobutane microbubbles) — The ultrasound contrast agent will be infused thorough an IV line and SHAPE ultrasound imaging and data acquisition will be performed with a Logiq E10 (GE Medical Systems, Waukesha, WI) ultrasound scanner.
  Arms: Longitudinal SHAPE; SHAPE with Sonazoid
Drug: SHAPE measurement using the ultrasound contrast agent Lumason (sulfur hexafluoride lipid-type A microspheres) — The ultrasound contrast agent will be infused thorough an IV line and SHAPE ultrasound imaging and data acquisition will be performed with a Logiq E10 (GE Medical Systems, Waukesha, WI) ultrasound scanner.
  Arms: Longitudinal SHAPE; SHAPE with Lumason

SUMMARY:
Early diagnosis of portal hypertension is difficult as symptoms rarely manifest until the later stages of liver disease. Both cirrhotic and non-cirrhotic portal hypertension can result in life-threatening complications, the most frequent of which is bleeding from esophageal varices. In children, variceal bleeds are associated with mortality rates of 1-3 %, while life-threatening complications have been reported in up to 20 % of children with cirrhosis. Despite the high incidence of portal hypertension in children with liver disease, a noninvasive modality to monitor disease progression and risk of complications is currently lacking. Hence, this trial will investigate the safety and efficacy of subharmonic aided pressure estimation (SHAPE) as a noninvasive ultrasound technique for diagnosing portal hypertension in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of chronic liver disease without portal hypertension.
* Patients with a diagnosis of chronic liver disease with portal hypertension.

Exclusion Criteria:

* Subjects who are pregnant.
* Patients with known or suspected hypersensitivity to egg phosphatidyl serine or with a history of anaphylactic allergy to eggs or egg products.
* Subjects with allergy to egg products or other components of the ultrasound contrast agents will be excluded.
* History of allergic reaction to Lumason®, sulfur hexafluoride, sulfur hexafluoride lipid microsphere components, or other ingredients in Lumason (polyethylene glycol, distearoylphosphatidylcholine (DSPC), dipalmitoylphosphatidylglycerol sodium (DPPG-Na), palmitic acid)
* History of allergic reaction to Sonazoid
* Patients with biliary atresia with asplenia or polysplenia.
* Patients with prior liver transplant.
* Patients with cystic fibrosis.
* Patients with chronic lung disease.
* Patients with portal vein thrombosis, cavernous transformation of the portal vein or absent portal vein.
* Adults not competent/impaired.
* Patients with significant heart disease or severe congenital heart disease

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The rate (%) of adverse events that occur with Sonazoid compared to the current rate of adverse events that have been reported in the Lumason package insert for pediatric use (0.001%) | 2 hours
Calibrated subharmonic microbubble signals (in dB) between the portal and hepatic veins will differentiate between the portal hypertension and non-portal hypertension groups with an accuracy of 94% | 2 hours

SECONDARY OUTCOMES:
Changes in calibrated subharmonic microbubble signals (in dB) between the portal and hepatic veins over time will predict the development of complications of portal hypertension (variceal bleeding, ascites, hepatopulmonary syndrome, etc) | on average 18 months
Calibrated subharmonic microbubble signals (in dB) between the portal and hepatic veins and liver fibrosis stage (on a scale from 0-4 as determined by liver biopsy) will correlate with a p<0.05 | 2 hours
Compare the calibrated subharmonic microbubble signals (in dB) between the portal and hepatic veins obtained with Lumason and Sonazoid, respectively, for their ability to differentiate between the portal hypertension and non-portal hypertension groups | 2 hours
Compare calibrated subharmonic microbubble signals (in dB) between the portal and hepatic veins to shear wave elastography values (in m/s) using regression analysis | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Forsberg, PhD, Principal Investigator — Thomas Jefferson University; Sudha A Anupindi, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated from the proposed study will be shared to make the results available to the scientific community.
  Presentations at national scientific meetings.
  Lectures.
  Post-graduate training.
  Approximately 12 months after the completion of the trial (when the main manuscript has been published) individual researchers can contact the PIs and request the final, complete data-set from this trial without any protected health information
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Approximately 12 months after the completion of the trial when the main manuscript has been published
Access Criteria: On an individual basis - contact the PIs

REFERENCES:
- [Background] Eisenbrey JR, Dave JK, Halldorsdottir VG, Merton DA, Miller C, Gonzalez JM, Machado P, Park S, Dianis S, Chalek CL, Kim CE, Baliff JP, Thomenius KE, Brown DB, Navarro V, Forsberg F. Chronic liver disease: noninvasive subharmonic aided pressure estimation of hepatic venous pressure gradient. Radiology. 2013 Aug;268(2):581-8. doi: 10.1148/radiol.13121769. Epub 2013 Mar 22. PMID 23525208
- [Background] Gupta I, Eisenbrey JR, Machado P, Stanczak M, Wessner CE, Shaw CM, Gummadi S, Fenkel JM, Tan A, Miller C, Parent J, Schultz S, Soulen MC, Sehgal CM, Wallace K, Forsberg F. Diagnosing Portal Hypertension with Noninvasive Subharmonic Pressure Estimates from a US Contrast Agent. Radiology. 2021 Jan;298(1):104-111. doi: 10.1148/radiol.2020202677. Epub 2020 Nov 17. PMID 33201789